CLINICAL TRIAL: NCT03845556
Title: Clinical Study of Titrating PEEP of Different Methods on Right Heart Function and Pulmonary Artery Pressure in ARDS Patients
Brief Title: Clinical Study of Titrating PEEP of Different Methods on Right Heart Function
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Southeast University, China (Other)
Collaborators: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Chun Pan, Clinical Professor, Southeast University, China
Other Study IDs: ARDS
Record Dates: First submitted 2018-10-11; First posted 2019-02-19 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: ARDS, Human
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To observe the influence of different methods titrating PEEP on right heart function and pulmonary artery pressure in ARDS patients .

DETAILED DESCRIPTION:
30 patients who diagnosed as ARDS were included in this study.Then set PEEP with respectively ARDS net 、EIT and Esophageal Pressure in Breathing Machine . Recorded diameter of right and left ventricular TAM TAPSE pulmonary artery pressure.Objective to evaluate the correlation between the level of PEEP in three methods and the right heart function and pulmonary artery pressure in ARDS patients .

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to ICU diagnosed of modecate to severe ARDS (Berlin criteria)
* Patients age between 18 years old and 80 years

Exclusion Criteria:

* Patients with chronic respiratory diseases such as COPD.
* Ventilated because of oesophageal surgery in the previous 12months.
* Patients who cannot obtain clear ultrasound images due to thoracic surgery ,massive pleural effusion.
* Oesophageal bleeding in previous 30 days history of oesophageal varices.
* Facial trauma and surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population admitted to ICU of Zhongda hospital，diagnosed of medium or serious ARDS。
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-08-04 (Actual); Primary Completion 2019-03-30 (Estimated); Study Completion 2019-03-30 (Estimated)

PRIMARY OUTCOMES:
the function of right heart and pulmonary artery pressure | 2018.4-2019.3
  Systolic Pulmonary Artery Pressure TAPSE or Tricuspid Annular Motion orTricuspid annular plane systolic excursion or right ventricular diameter or right left ventricular diameter ratio in diffrient PEEP

CONTACTS AND LOCATIONS:
Overall Officials: Chun Pan, Dr, Principal Investigator — southeast university
Locations (1):
- Zhongda Hospital, Nanjing, Jiangsu, China